CLINICAL TRIAL: NCT03901287
Title: Quantitative Dual Energy Computed Tomography in Pulmonary Hypertension "DECTPH".
Brief Title: Quantitative Dual Energy Computed Tomography in Pulmonary Hypertension
Acronym: DECTPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2018/59
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Pulmonary Hypertension
Keywords: pulmonary hypertension; dual energy CT; quantification; lung perfusion; prediction
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dual energy CT (Experimental): The procedure involves post processing and analysis of reconstructed images from dual energy CT scans available at the Bordeaux University Hospital and used in routine care, which will allow us to collect morphometric data (bronchial wall thickness and cross sectional area of small pulmonary vessels) and to assess pulmonary perfusion by studying iodine mapping and quantifying pulmonary perfusion blood volume (PVB)
  Interventions: Other: dual energy CT scans

INTERVENTIONS:
Other: dual energy CT scans — The procedure involves post processing and analysis of reconstructed images from dual energy CT scans available at the Bordeaux University Hospital and used in routine care, which will allow us to collect morphometric data (bronchial wall thickness and cross sectional area of small pulmonary vessels) and to assess pulmonary perfusion by studying iodine mapping and quantifying pulmonary perfusion blood volume (PVB)

SUMMARY:
Pathophysiological mechanisms leading to pulmonary hypertension (PH) are complex. Quantitative computed tomography (QCT) can help us to study morphological alterations in patients with PH. These CT morphometrics are useful to predict the degree of PH severity at least in PH secondary to chronic obstructive pulmonary disease (COPD). We hypothesized that assessing lung perfusion using dual energy CT (DECT) can refine our knowledge on PH pathophysiology and help to predict PH severity irrespective of its etiology

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) is a serious disease with poor prognosis and high morbidity and mortality. It is defined as an increase in mean pulmonary arterial pressure (mPAP) above or equal to 25 mmHg measured by right heart catheterization, which is an invasive technique.

Computed tomography (CT) plays an important role in the classification of PH and the identification of pulmonary etiologies responsible for PH (chronic obstructive pulmonary disease (COPD), idiopathic pulmonary fibrosis...) or signs of chronic thromboembolic PH (CTEPH).

Quantitative CT allows accurate analysis of the morphological changes found in PH and leading to a better understanding of the complex interactions involved (arterial and bronchial remodeling in PH secondary to COPD, inflammation etc.).

Dual energy CT acquisition has shown its interest in helping to diagnose pulmonary embolism. It provides information on pulmonary perfusion by performing iodine mapping and measuring pulmonary perfusion blood volume (PVB).

This project intends to study morphological and functional alterations at bronchial and vascular levels in PH patients using quantitative DECT and to examine their impact to predict existence and severity of PH irrespective of its etiology. To measure from DECT scan images, cross sectional area of small pulmonary vessels (CSA), bronchial wall thickness (WT) and pulmonary perfusion blood volume. To collect data from right heart catheterization, echocardiography, pulmonary functional tests and blood tests. All these examinations will be performed in routine care within a week after the patient is referred to our institution. Statistical analysis of these parameters could lead to a multivariate model able to predict existence and severity of PH.

In addition, DECT allows the use of low energy (low Kilovoltage), which increases contrast and improves segmentation of the pulmonary arteries. Thus, peripheral pulmonary arteries and veins can be distinguishable in order to evaluate not just the sectional area of the small pulmonary vessels but also 3D volume of small pulmonary arteries (VSA). This technical modification would make it possible to refine the quantitative exploration of the vascular compartment of PH

ELIGIBILITY:
Inclusion Criteria:

* adults (18 years old and over)
* Patient with PH diagnosed at right heart catheterization
* Availability of a dual energy chest CT scans with contrast injection performed as part of standard patient workup
* Patient's consent or authorisation for data processing.

Exclusion Criteria:

* patient without any chest CT scan available or planned in the patient workup

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
stence and the severity of PH | Baseline
  Prediction of the existence and the severity of PH using a qCT score combining morphometric parameters (WT(mm), CSA(mm2) and/or VSA(mm3)) and functional parameters (PVB(HU))

SECONDARY OUTCOMES:
kappa coefficient | baseline
  Good kappa coefficient (>0.6) for topographic evaluation of pulmonary artery segmentation
Dice coefficient | Baseline
  Good Dice coefficient (>0.8) for overlap and similarity between manual (ground truth) and automatic segmentations

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No